CLINICAL TRIAL: NCT02224300
Title: Nursing Care With Patients With Venous Leg Ulcers - Developing an Internet-based Education Program and Evaluation of Its Effectiveness
Brief Title: Nursing Care With Patients With Venous Leg Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Minna Ylönen, PhD candidate, University of Turku
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LAPHOI
Record Dates: First submitted 2014-08-09; First posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: - Venous Leg Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Education (Experimental): Intervention group will receive the ELC for six weeks (15.9. - 26.10.2014) and comparison group will not receive it.
  Members of the intervention group in will work in teams of 10 nurses with weekly questions (released in Mondays) based on patient-description existing in Moodle. One member of the team will send the solutions to questions once a week (in Thursdays) Moodle. Researcher will download the model-answer to Moodle once a week (in Fridays) and nurses will compare their answer to model answer (self-evaluation).
  Interventions: Behavioral: Internet-based education of venous leg ulcer nursing care

INTERVENTIONS:
Behavioral: Internet-based education of venous leg ulcer nursing care — Intervention is delivering the ELC (Electronic Learning of venous leg ulcer nursing care) to home health-care nurses (registered nurses, public health nurses and licensed practical nurses) . The ELC development was based on the integrative literature review about nurses' knowledge gaps on venous leg ulcer nursing care. The pedagogical basis of the ELC is constructivism and blended learning approach. The ELC comprises contact learning and distance learning. Content of ELC is evidence-based information already existing in Internet and the basis of the information is the Finnish Current Care Guidelines for Chronic leg ulcers (2014), which are evidence-based clinical practice guidelines. They are intended as basis for ulcer treatment decisions, and guidelines can be used by nurses and other healthcare professionals.

SUMMARY:
Aims are:

* develop an Internet-based education programme about venous leg ulcer nursing care (ELC)
* evaluate the clinical, cognitive and economical outcomes of education programme

Research questions are:

1. What are the cognitive outcomes of ELC (perceived knowledge, attitudes towards venous leg ulcer nursing care, theoretical knowledge level and practical knowledge)?

Hypotheses for research question 1 are:

1. Nurses using the ELC will have better knowledge (perceived, practical and theoretical knowledge) than those who will not use the ELC.
2. Nurses using the ELC will have more positive attitudes towards venous leg ulcer nursing care than those who will not use the ELC.

2. What are the clinical outcomes of ELC (ulcer healing, ulcer size, treatment supplies)?

Hypotheses for research question 2 are:

1. Ulcer healing progresses better among patients who are taken care by nurses using the ELC.
2. Ulcer sizes will be 10 % smaller among the patients cared for nurses using the ELC.
3. Nurses using the ELC will use mire adequate treatment supplies than those who will not use the ELC.

3. What are the economical outcomes (treatment time and supply usage) of ELC?

Hypothesis for research question 3 is:

1. The economical expenditures will be lower among nurses using the ELC.

The ultimate aim is to promote evidence-based nursing care among patients with venous leg ulcer.

DETAILED DESCRIPTION:
The study takes place in home-care in two Finnish municipality, which are similar size and staff structure and working ideology are basically the same.

Enrolment of participants has started with information occasion in both municipalities in June 2014. Nurses were asked to fill the Patients Clinical Situation Questionnaire, handouts and forms for informed consent were delivered. (Figure 1) All eligible nurses and patients will be identified with Patient Clinical Assessment. The sample size was determined with power analysis and the result was that 200 nurses are needed in the intervention group and 100 nurses in the comparison group.

ELIGIBILITY:
Inclusion criteria for nurses:

1. Working in municipality home-care
2. Permanent attachment or three months or longer temporary post in municipality home-care
3. Working in home-care area where patients with chronic leg ulcer are taken care during the study

Exclusion criteria for nurses:

1. Working in other place than home-care There are no other exclusion criteria.

Inclusion criteria for patients to observation are:

1. Home health-care patient aged 60 or over
2. Venous leg ulcer diagnosis
3. Chronic ulcer in the lower leg without diagnosis

Exclusion criteria for patients:

1. An ulcer with other diagnosis than venous leg ulcer diagnosis There are no other exclusion criteria for patients.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Changes in nurses´ knowledge before and after the education | Baseline, Week 8 and Week 12
  Knowledge is divided into nurses´ perceived knowledge, practical and theoretical knowledge.
  Changes in perceived knowledge will be measured with structured self-completed questionnaire.
  Changes in practical knowledge will be measured with structured observation. Changes in theoretical knowledge will be measured with structured questionnaire (knowledge-test).

SECONDARY OUTCOMES:
Changes in nurses´ attitudes towards patients with venous leg ulcers before and after the education | Baseline, Week 8 and Week 12
  Changes in attitudes will be measured with structured questionnaire.
Changes in clinical variables; venous leg ulcer size. | Baseline, Week 8 and Week 12
  Changes in venous leg sizes variables will be measured during observations. Each venous leg ulcer will measured with paper ruler.
Changes in clinical variables; adequacy of the supplies used. | Baseline, Week 8 and Week 12
  Changes in adequacy of supplies used will be measured with structured observation.
Changes in economical variables cost of supplies and treatment time. | Baseline, Week 8 and Week 12
  Changes in economical variables will be measured with structured observation.

CONTACTS AND LOCATIONS:
Locations (1):
- Homecare, Turku, Finland

REFERENCES:
- [Derived] Ylonen M, Viljamaa J, Isoaho H, Junttila K, Leino-Kilpi H, Suhonen R. Effectiveness of an Internet-based learning program on venous leg ulcer nursing care in home health care--study protocol. J Adv Nurs. 2015 Oct;71(10):2413-25. doi: 10.1111/jan.12683. Epub 2015 May 14. PMID 25976713